CLINICAL TRIAL: NCT00485147
Title: Study of Human Locomotion With Global Positioning System. Application to Patients With Peripheral Arterial Disease
Brief Title: Locomotion and Global Positioning System in Arterial Disease
Acronym: Starter-GPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Société Française de Médecine Vasculaire (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CP 2005-04
Record Dates: First submitted 2007-06-11; First posted 2007-06-12 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2010-04

CONDITIONS: Peripheral Arterial Disease
Keywords: Claudication; peripheral arterial disease; Diagnosis; Exercise; Walking impairment; Disability
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Disease; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Recording of GPS during a free walking in a public park — Analyse the clinical change after surgery from GPS measurements and compare it with laboratory measurement.

SUMMARY:
The maximal walking distance (MWD) performed on treadmill (TT) remains the gold standard in estimating the walking capacity of patients suffering from peripheral arterial disease (PAD) with intermittent claudication, although treadmills are not accessible to most physicians. We hypothesized that global positioning system (GPS) recordings could monitor community-based outdoor walking and provide valid information on walking capacity in PAD patients.

DETAILED DESCRIPTION:
The study has two main objectives, conducted together. Each objective include several phases.

Objective 1: technical validation of GPS measurements in healthy subjects.

phase 1: technical validation of a GPS device to study outdoor walking (completed).

phase 2: comparison and use of various GPS devices (intra- and inter-GPS variability) in the study outdoor walking (on-going).

phase 3: study of several factors that could influence accuracy of GPS measurements as walking speed, environment, sampling frequency and others technical features as the WAAS/EGNOS function (on-going).

Objective 2: Application in PAD patients to study walking capacity under free-living conditions

phase 1: comparison of GPS measurements (maximal walking distance) with the gold standard treadmill measurement of maximal walking distance (completed).

phase 2: analysis of the variability of the walking capacity under free-living conditions from GPS measurements (completed).

phase 3: study of reliability and sensibility (effect of treatment) of GPS measurements (on-going).

phase 4: study of the relationship between laboratory measurements of walking capacity and GPS-derived parameters.

ELIGIBILITY:
Inclusion Criteria:

* Ankle to Brachial Index (ABI) < 0.95 for PAD patients
* Age > 18 years old
* Able to walk on treadmill

Exclusion Criteria:

* limb pain of potential non-vascular origin
* myocardial infraction in the last six months
* uncontrolled angina pectoris

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2006-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Validate the ability of GPS to detect walking and resting bouts and to accurately estimate walking speed and distance in normal subjects. | 2 years
Measurement of maximal walking distance using GPS and comparison with treadmill measurement in PAD patients. | 2 years

SECONDARY OUTCOMES:
Determine the variability of the walking capacity and its potential determinants in PAD patients. | 3 years
Analyse the reliability and sensibility of GPS measurements of the walking capacity in PAD patients. | 4 years
Analyse potential factors that could affect the accuracy of GPS measurements | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Abraham, MD, PhD, Study Director — Laboratory for Vascular Investigations. University Hospital. Angers. France.
Locations (1):
- Centre hospitalier universitaire, Angers, France

REFERENCES:
- [Derived] Noury-Desvaux B, Abraham P, Mahe G, Sauvaget T, Leftheriotis G, Le Faucheur A. The accuracy of a simple, low-cost GPS data logger/receiver to study outdoor human walking in view of health and clinical studies. PLoS One. 2011;6(9):e23027. doi: 10.1371/journal.pone.0023027. Epub 2011 Sep 13. PMID 21931593
- [Derived] Le Faucheur A, Noury-Desvaux B, Mahe G, Sauvaget T, Saumet JL, Leftheriotis G, Abraham P. Variability and short-term determinants of walking capacity in patients with intermittent claudication. J Vasc Surg. 2010 Apr;51(4):886-92. doi: 10.1016/j.jvs.2009.10.120. PMID 20347684